CLINICAL TRIAL: NCT03997006
Title: Is Aminophylline More Effective Than Neostigmine/Atropine Mixture in the Treatment of Post-dural Puncture Headache: A Randomized Clinical Trial
Brief Title: Is Aminophylline More Effective Than Neostigmine/Atropine Mixture in the Treatment of Post-dural Puncture Headache
Acronym: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DTH:19001
Record Dates: First submitted 2019-06-20; First posted 2019-06-25 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Post-Dural Puncture Headache
Keywords: Aminophylline; Atropine; Neostigmine; Post-dural puncture headache; Spinal anesthesia
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Aminophylline; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (n=30) (Active Comparator): Aminophylline group
  Interventions: Drug: IV Aminophylline
- Group NA (n=30) (Active Comparator): Neostigmine/Atropine group
  Interventions: Drug: IV Neostigmine Methylsulfate + Atropine Sulphate

INTERVENTIONS:
Drug: IV Aminophylline — IV Aminophylline (100 mg/8h)
  Other Names: Minophylline-N ampoule
  Arms: Group A (n=30)
Drug: IV Neostigmine Methylsulfate + Atropine Sulphate — IV Neostigmine/Atropine mixture (20 μg/kg Neostigmine + 10 μg/kg Atropine)/8h
  Other Names: Neostigmine ampoule, Atropine ampoule
  Arms: Group NA (n=30)

SUMMARY:
Objectives: To compare the safety and efficacy of IV aminophylline versus IV neostigmine/atropine mixture in the treatment of post-dural puncture headache (PDPH).

Background: PDPH is the most frequent complication of procedures associated with dural puncture for spinal anesthesia or following accidental dural puncture during epidural anesthesia. Since invasive treatments have known complications, pharmacologic management may be preferable.

Patients and Methods: This was a prospective, randomized, double-blind, phase four clinical trial; carried out on 60 patients presented with PDPH at our hospital. Patients were randomly allocated into two equal groups (30 patients each); group A, received IV aminophylline, and group NA, received IV neostigmine/atropine mixture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NPRS score of ≥ 5
* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 50 years

Exclusion Criteria:

* Patients with NPRS score < 5
* ASA physical status > II
* Age < 21 years or > 50 years
* Pregnant women
* History of; chronic headache, Cluster headache, Migraine
* History of; Convulsions, Cerebrovascular accident, Previous neurological diseases
* Signs of meningismus
* Bronchial asthma
* Arrhythmia
* Hypertension
* Ischemic heart disease
* Hyperthyroidism

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Median and Range of Numeric Pain Rating Scale (NPRS) score | 48 hours after initiation of treatment
  NPRS measures the severity of PDPH, it is a 11 point scale from 0-10; where 0=No pain and 10=Worst possible pain (before, 2h, 6h, 12h, then every 12h till 48h)

SECONDARY OUTCOMES:
Mean and Standard deviation of PDPH duration (hours) (mean±SD) | 48 hours after initiation of treatment
  Time from PDPH onset till NPRS score ≤ 3
Number of participants and Rate of Treatment-related complications | 48 hours after initiation of treatment
  Number of participants and Rate of: Diarrhea, Palpitation, Abdominal cramps, Muscle twitches, Bronchospasm, Urinary bladder hyperactivity

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt